CLINICAL TRIAL: NCT00415766
Title: Recombinant hCG (Ovitrelle) Vesrus Urinary hCG (Pregnyl) for Triggering Final Oocyte Maturation in High Responders
Brief Title: Comparison Between Recombinant Versus Urinary hCG for Ovulation Induction in High Responders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ovitrelle vs pregnyl
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: recombinant hCG; urinary hCG
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- rHCG 250 ug (Active Comparator): Injection of 250 ug Ovitrelle to trigger final oocyte maturation
  Interventions: Drug: rHCG 250ug
- uHCG 5000 IU (Active Comparator): Injection of 5000 IU Pregnyl to trigger final oocyte maturation
  Interventions: Drug: uHCG 5000 IU
- uHCG 7500 IU (Active Comparator): Injection of 7500 IU Pregnyl to trigger final oocyte maturation
  Interventions: Drug: uHCG 7500 IU

INTERVENTIONS:
Drug: rHCG 250ug — Injection of 250 ug Ovitrelle to trigger final oocyte maturation
  Other Names: Ovitrelle
  Arms: rHCG 250 ug
Drug: uHCG 5000 IU — Injection of 5000 IU Pregnyl to trigger final oocyte maturation
  Other Names: Pregnyl 5000 IU
  Arms: uHCG 5000 IU
Drug: uHCG 7500 IU — Injection of 7500 IU Pregnyl to trigger final oocyte maturation
  Other Names: Pregnyl 7500 IU
  Arms: uHCG 7500 IU

SUMMARY:
The purpose of this study is to compare the clinical outcomes of recombinant human chorionic gonadotrophin (rHCG) and urinary HCG (uHCG) in patients undergoing IVF cycles.

DETAILED DESCRIPTION:
Urinary human chorionic gonadotrophin (u-hCG) has been widely used to induce final oocyte maturation and to trigger ovulation in assisted conception. Recombinant technology has allowed the production of r-hCG inj which all urinary contaminants are absent. Hence, this would allow the safe subcutaneous administration of a compound with less batch-to-batch variation. This study will investigate the effectiveness of the recombinant hCG compared to the currently used urinary hCG.

ELIGIBILITY:
Inclusion Criteria:

* At least 14 follicles >11mm on the day of triggering final oocyte maturation
* Pretreated with GnRH antagonist protocol

Exclusion Criteria:

* Poor responders
* Women with 25 or more follicles on the day of trigger

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of mature oocytes | Day of oocyte retrieval (Day 0)
  Percentage MII/COCs

SECONDARY OUTCOMES:
Positive test per embryo transfer | 15 days post oocyte retrieval
Clinical pregnancy per embryo transfer | 7 weeks of gestation
Ongoing pregnancy per embryo transfer | 12 weeks of gestation
Level of serum hCG on day of oocyte retrieval | Day of oocyte retrieval
Number of oocytes (COC) retrieved | Day of oocyte retrieval
Number of mature oocytes (MII) | Day of oocyte retrieval
Oocyte retrieval rate | Day of oocyte retrieval (Day 0)
  Number of oocytes retrieved/number of follicles on the day of triggering final oocyte maturation
Incidence of severe early OHSS | up to Day 5 post oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia, Athens, Greece

REFERENCES:
- [Background] Revelli A, Poso F, Gennarelli G, Moffa F, Grassi G, Massobrio M. Recombinant versus highly-purified, urinary follicle-stimulating hormone (r-FSH vs. HP-uFSH) in ovulation induction: a prospective, randomized study with cost-minimization analysis. Reprod Biol Endocrinol. 2006 Jul 18;4:38. doi: 10.1186/1477-7827-4-38. PMID 16848893
- [Background] Al-Inany HG, Aboulghar M, Mansour R, Proctor M. Recombinant versus urinary human chorionic gonadotrophin for ovulation induction in assisted conception. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003719. doi: 10.1002/14651858.CD003719.pub2. PMID 15846677